CLINICAL TRIAL: NCT06995079
Title: Comparison of the Effects of Pericapsular Nerve Group Block (Peng Block) and Lumbar Erector Spinae Plane Block (Lesp Block) on Postoperative Opioid Consumption in Geriatric Patients Undergoing Hip Fracture Surgery
Brief Title: Comparıson Of The Effects Of Perıcapsulary Nerve Group Block (Peng Block) And Lumbar Erector Spına Plan Block (Lesp Block) On Postoperatıve Opıoıd Consumptıon
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PENGVSLESP
Record Dates: First submitted 2025-05-07; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Pengblock; over65years; Lumbar Erector Spinae Plane Block; Hipfracture

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pericapsular nerve group block (peng block) (Experimental): The patient will first be taken to the block room in the operating room.In this group, patients will be given a Peng block before surgery.The patient will then be taken to the operating room and spinal anesthesia will be applied.Postoperative analgesia requirement will be assessed
  Interventions: Procedure: Postoperative pain assessment of patients who underwent block
- lumbar erector spinae plane block(lesp block) (Experimental): The patient will first be taken to the block room in the operating room.In this group, patients will be given a lumbar erector spinae plane block before surgery.The patient will then be taken to the operating room and spinal anesthesia will be applied.Postoperative analgesia requirement will be assessed
  Interventions: Procedure: Postoperative pain assessment of patients who underwent block

INTERVENTIONS:
Procedure: Postoperative pain assessment of patients who underwent block — Postoperative pain assessment of patients who underwent block

SUMMARY:
The aim is to demonstrate that lumbar ESP block provides more effective postoperative analgesia than PENG block in geriatric patients with hip fractures, and reduces postoperative opioid consumption more than PENG block

ELIGIBILITY:
Inclusion Criteria:

* patients with hip fractures
* over 65 years old

Exclusion Criteria:

* long-term surgery
* Patients who do not want regional anesthesia
* bleeding disorder disease
* wound in the operation area

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 6 month
  To evaluate postoperative pain after two different block applications in patients undergoing hip fracture surgery.Evaluation of patients' postoperative 30th minute, 2nd hour, 6th hour, 12th hour and 24th hour verbal analog scores.To examine the total fentanyl consumption, acetaminophen consumption, and nonsteroidal anti-inflammatory drug consumption of patients in the postoperative 24 hours.